CLINICAL TRIAL: NCT07057570
Title: Comparison of Pre Existing Intra Operative Thyroidectomy Difficulty Score With Novel Difficult Thyroidectomy Predictor Score in Prediction of Difficult Thyroidectomies
Acronym: Thyroid Score
Status: Completed | Type: Observational
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Umaiya/Kemu
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Thyroidectomy; Thyroid Gland Disease
Keywords: Difficult thyroidectomies; TDS score
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients undergoing thyroidectomy: No intervention , just observation

SUMMARY:
Novel Difficult Thyroidectomy Score to predict Difficult thyroidectomies pre operatively .

DETAILED DESCRIPTION:
A newer score has been formulated that will help to predict the level of difficulty that surgeon may encouter during any thyroidectomy unlike before where there was no such tool and only intra operatively surgeon realized he has opened a very difficult thyroid case.

ELIGIBILITY:
Inclusion Criteria:

* All MNG undergoing thyroidectomy Euthyroid /toxic controlled cases Age 18-60yrs Both genders

Exclusion Criteria:

* carcinomas Co morbs Toxicity signs Pregnancy /lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pakistani Local population (Asian)
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Difficult thyroidectomy | Time required for surgery
  Any thyroidectomy with score cut off value > 10

CONTACTS AND LOCATIONS:
Locations (1):
- Kemu, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Not sure how and why i should share my IPD with others